CLINICAL TRIAL: NCT00109343
Title: An Open, Randomized, Multicenter Study of the Safety, Tolerability, and Immunogenicity of V221 Given Concomitantly With Pneumococcal Conjugate Vaccine in Healthy Children 12 to 15 Months of Age
Brief Title: V221 Concomitant Use Study With Pneumococcal Conjugate Vaccine (V221-019)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V221-019; 2005_027
Record Dates: First submitted 2005-04-27; First posted 2005-04-27 (Estimated); Results first posted 2010-02-10 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Measles; Mumps; Rubella; Varicella
MeSH Terms: conditions — Measles; Mumps; Rubella; Chickenpox | interventions — measles, mumps, rubella, varicella vaccine; Pneumococcal Vaccines; Heptavalent Pneumococcal Conjugate Vaccine

ARMS (3):
- 1 (Experimental): Group 1: ProQuad™ (V221) + PREVNAR™ (pneumococcal 7-valent conjugate vaccine) followed by ProQuad™ (Day 91)
  Interventions: Biological: Comparator: ProQuad™ (V221); Biological: Comparator: PREVNAR™ (pneumococcal 7-valent conjugate vaccine)
- 2 (Experimental): Group 2: PREVNAR™ followed by ProQuad™ (Day 43) followed by ProQuad™ (Day 133)
  Interventions: Biological: Comparator: ProQuad™ (V221); Biological: Comparator: PREVNAR™ (pneumococcal 7-valent conjugate vaccine)
- 3 (Experimental): Group 3: ProQuad™ followed by PREVNAR™ (Day 43), followed by ProQuad™ (Day 91)
  Interventions: Biological: Comparator: ProQuad™ (V221); Biological: Comparator: PREVNAR™ (pneumococcal 7-valent conjugate vaccine)

INTERVENTIONS:
Biological: Comparator: ProQuad™ (V221) — 0.5-mL subcutaneous injection of measles, mumps, rubella, varicella virus vaccine live (MMRV)
  Other Names: ProQuad™; V221
Biological: Comparator: PREVNAR™ (pneumococcal 7-valent conjugate vaccine) — 0.5-mL intramuscular injection of pneumococcal 7-valent conjugate vaccine
  Other Names: PREVNAR™

SUMMARY:
The study is being conducted to demonstrate that V221 may be administered concomitantly with pneumococcal conjugate vaccine without impairing the safety or immunogenicity of measles, mumps, rubella, varicella, or the 7 serotypes of S. pneumoniae.

ELIGIBILITY:
Inclusion Criteria:

* In good health
* 12 to 15 months of age
* Negative clinical history to measles, mumps, rubella, varicella and/or zoster
* Received only the 3-dose primary series of a pneumococcal conjugate vaccine with at least 2 months prior to the receipt of any of the study vaccines
* Signed consent

Exclusion Criteria:

* Previous administration of any measles, mumps, rubella, or varicella vaccine either alone or in any combination
* Any condition resulting in depressed immunity
* Any allergy to any vaccine component as stated in the package circulars
* Exposure to measles, mumps, rubella, varicella, or zoster within 4 weeks prior to the study vaccination
* History of seizure disorder
* Receipt of an inactivated vaccine within 14 days prior to enrollment or live vaccine within 30 days
* Recent febrile illness

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1027 (Actual)
Dates: Start 2006-03; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Leonardi M, Bromberg K, Baxter R, Gardner JL, Klopfer S, Nicholson O, Brockley M, Trammel J, Leamy V, Williams W, Kuter B, Schodel F. Immunogenicity and safety of MMRV and PCV-7 administered concomitantly in healthy children. Pediatrics. 2011 Dec;128(6):e1387-94. doi: 10.1542/peds.2010-2132. Epub 2011 Nov 28. PMID 22123890

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 clinical sites in the United States
  Date first participant visit: 06-Mar-2006
  Date last participant visit: 14-Sep-2007
Groups:
- Group 1 - ProQuad™ + PREVNAR™: Group 1 - ProQuad™ (measles, mumps, rubella, and varicella vaccine) + fourth dose of PREVNAR™ (pneumococcal 7-valent conjugate vaccine) administered concomitantly at separate injection sites on Day 1. Second dose of ProQuad™ administered at least 90 days (Day 91) after the first dose.
- Group 2 - PREVNAR™ Followed by ProQuad™: Group 2 - Fourth dose of PREVNAR™ (pneumococcal 7-valent conjugate vaccine) administered on Day 1. ProQuad™ (measles, mumps, rubella, and varicella vaccine) administered on Day 43. Second dose of ProQuad™ administered at least 90 days (Day 133) after the first dose.
- Group 3 - ProQuad™ Followed by PREVNAR™: Group 3 - ProQuad™ (measles, mumps, rubella, and varicella vaccine) administered on Day 1. Fourth dose of PREVNAR™ (pneumococcal 7-valent conjugate vaccine) administered on Day 43. Second dose of ProQuad™ administered at least 90 days (Day 91) after the first dose.
Period: Overall Study
Arm/Group | Group 1 - ProQuad™ + PREVNAR™ | Group 2 - PREVNAR™ Followed by ProQuad™ | Group 3 - ProQuad™ Followed by PREVNAR™
Started | 510 | 258 | 259
Vaccinated at Visit 1 | 510 | 258 | 259
Vaccinated at Visit 2 | 0 (Per-protocol, subjects in Group 1 were not vaccinated at Visit 2) | 246 | 246
Vaccinated at Visit 4 | 466 | 235 | 240
Completed | 446 | 221 | 229
Not Completed | 64 | 37 | 30
Not completed — Adverse Event | 1 | 0 | 2
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Lost to Follow-up | 35 | 20 | 14
Not completed — Protocol Violation | 1 | 2 | 2
Not completed — Withdrawal by Subject | 15 | 11 | 10
Not completed — Subject Moved | 6 | 2 | 1
Not completed — Other | 5 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - ProQuad™ + PREVNAR™ | Group 2 - PREVNAR™ Followed by ProQuad™ | Group 3 - ProQuad™ Followed by PREVNAR™ | Total
Number analyzed (Participants) | 510 | 258 | 259 | 1027
Age, Continuous [Mean (Standard Deviation); unit: Months] | 12.6 (0.96) | 12.5 (0.93) | 12.6 (0.98) | 12.6 (0.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 230 | 120 | 117 | 467
  Male | 280 | 138 | 142 | 560
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 18 | 5 | 8 | 31
  Black | 83 | 36 | 36 | 155
  Hispanic | 46 | 31 | 26 | 103
  White | 335 | 161 | 174 | 670
  Other | 28 | 25 | 15 | 68

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postvaccination Measles Enzyme-Linked Immunosorbent Assay (ELISA) Antibody Titer ≥255 mIU/mL
Description: Antibody Response to Measles at 6 Weeks Postvaccination for Subjects Initially Seronegative (a titer <255 mIU/mL) to Measles at Baseline.
Time Frame: 6 weeks Postvaccination in subjects receiving ProQuad™ concomitantly with a fourth dose of Prevnar™ and in subjects receiving ProQuad™ alone
Population: Per-protocol analysis set includes participants who had pre- and postvaccination blood samples within predefined day ranges, were seronegative to measles at baseline, and followed protocol procedures.
Measure: Number; unit: Participants
Arm/Group | Group 1 - ProQuad™ + PREVNAR™ | Group 3 - ProQuad™ Followed by PREVNAR™
Number analyzed (Participants) | 406 | 204
Participants | 395 | 203

2. Primary Outcome: Number of Participants With Postvaccination Mumps ELISA Antibody Titer ≥10 Ab Units/mL
Description: Antibody Response to Mumps at 6 Weeks Postvaccination for Subjects Initially Seronegative (a titer <10 ELISA Ab units/mL) to Mumps at Baseline.
Time Frame: as for outcome 1
Population: Per-protocol analysis set includes participants who had pre- and postvaccination blood samples within predefined day ranges, were seronegative to mumps at baseline, and followed protocol procedures.
Measure: Number; unit: Participants
Arm/Group | Group 1 - ProQuad™ + PREVNAR™ | Group 3 - ProQuad™ Followed by PREVNAR™
Number analyzed (Participants) | 403 | 208
Participants | 390 | 205

3. Primary Outcome: Number of Participants With Postvaccination Rubella ELISA Antibody Titer ≥10 IU/mL
Description: Antibody Response to Rubella at 6 Weeks Postvaccination for Subjects Initially Seronegative (a titer <10 IU/mL) to Rubella at Baseline.
Time Frame: as for outcome 1
Population: Per-protocol analysis set includes participants who had pre- and postvaccination blood samples within predefined day ranges, were seronegative to rubella at baseline, and followed protocol procedures.
Measure: Number; unit: Participants
Arm/Group | Group 1 - ProQuad™ + PREVNAR™ | Group 3 - ProQuad™ Followed by PREVNAR™
Number analyzed (Participants) | 377 | 195
Participants | 372 | 191

4. Primary Outcome: Number of Participants With Postvaccination Varicella Antibody Titer ≥1.25 Glycoprotein Enzyme-Linked Immunosorbent Assay (gpELISA) Units/mL and ≥5 gpELISA Units/mL
Description: Antibody Response to Varicella at 6 Weeks Postvaccination for Subjects Initially With Varicella Antibody Titer <1.25 gpELISA units/mL at Baseline
Time Frame: as for outcome 1
Population: Per-protocol analysis set includes participants who had pre- and postvaccination blood samples within predefined day ranges, Varicella Antibody Titer <1.25 gpELISA units/mL at baseline, and followed protocol procedures.
Measure: Number; unit: Participants
Arm/Group | Group 1 - ProQuad™ + PREVNAR™ | Group 3 - ProQuad™ Followed by PREVNAR™
Number analyzed (Participants) | 379 | 192
Participants
  Number of Participants ≥1.25 gpELISA units/mL | 374 | 187
  Number of Participants ≥5 gpELISA units/mL | 350 | 169

5. Other Pre Specified Outcome: Number of Participants With Postvaccination Pneumococcal Polysaccharide ELISA Titer ≥0.2 mcg/mL for S. Pneumoniae Serotype 4
Time Frame: 6 weeks Postvaccination in subjects receiving ProQuad™ concomitantly with a fourth dose of Prevnar™ and in subjects receiving a fourth dose of Prevnar™ alone
Population: Per-protocol analysis set includes participants who had pre- and postvaccination blood samples within predefined day ranges and followed protocol procedures.
Measure: Number; unit: Participants
Arm/Group | Group 1 - ProQuad™ + PREVNAR™ | Group 2 - PREVNAR™ Followed by ProQuad™
Number analyzed (Participants) | 410 | 193
Participants | 403 | 193

6. Other Pre Specified Outcome: Number of Participants With Postvaccination Pneumococcal Polysaccharide ELISA Titer ≥0.2 mcg/mL for S. Pneumoniae Serotype 6B
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Group 1 - ProQuad™ + PREVNAR™ | Group 2 - PREVNAR™ Followed by ProQuad™
Number analyzed (Participants) | 410 | 192
Participants | 408 | 192

7. Other Pre Specified Outcome: Number of Participants With Postvaccination Pneumococcal Polysaccharide ELISA Titer ≥0.2 mcg/mL for S. Pneumoniae Serotype 9V
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Group 1 - ProQuad™ + PREVNAR™ | Group 2 - PREVNAR™ Followed by ProQuad™
Number analyzed (Participants) | 409 | 193
Participants | 407 | 193

8. Other Pre Specified Outcome: Number of Participants With Postvaccination Pneumococcal Polysaccharide ELISA Titer ≥0.2 mcg/mL for S. Pneumoniae Serotype 14
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Group 1 - ProQuad™ + PREVNAR™ | Group 2 - PREVNAR™ Followed by ProQuad™
Number analyzed (Participants) | 408 | 193
Participants | 407 | 193

9. Other Pre Specified Outcome: Number of Participants With Postvaccination Pneumococcal Polysaccharide ELISA Titer ≥0.2 mcg/mL for S. Pneumoniae Serotype 18C
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Group 1 - ProQuad™ + PREVNAR™ | Group 2 - PREVNAR™ Followed by ProQuad™
Number analyzed (Participants) | 408 | 193
Participants | 404 | 191

10. Other Pre Specified Outcome: Number of Participants With Postvaccination Pneumococcal Polysaccharide ELISA Titer ≥0.2 mcg/mL for S. Pneumoniae Serotype 19F
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Group 1 - ProQuad™ + PREVNAR™ | Group 2 - PREVNAR™ Followed by ProQuad™
Number analyzed (Participants) | 408 | 192
Participants | 407 | 192

11. Other Pre Specified Outcome: Number of Participants With Postvaccination Pneumococcal Polysaccharide ELISA Titer ≥0.2 mcg/mL for S. Pneumoniae Serotype 23F
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Group 1 - ProQuad™ + PREVNAR™ | Group 2 - PREVNAR™ Followed by ProQuad™
Number analyzed (Participants) | 413 | 197
Participants | 412 | 194

12. Primary Outcome: Antibody Response to S. Pneumoniae Serotype 4 - Geometric Mean Titer
Description: Postvaccination observed Geometric Mean Titer of antibody to S. Pneumoniae serotype 4
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Group 1 - ProQuad™ + PREVNAR™ | Group 2 - PREVNAR™ Followed by ProQuad™
Number analyzed (Participants) | 410 | 193
mcg/mL | 1.54 [1.41 to 1.67] | 1.34 [1.19 to 1.51]

13. Primary Outcome: Antibody Response to S. Pneumoniae Serotype 6B - Geometric Mean Titer
Description: Postvaccination observed Geometric Mean Titer of antibody to S. Pneumoniae serotype 6B
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Group 1 - ProQuad™ + PREVNAR™ | Group 2 - PREVNAR™ Followed by ProQuad™
Number analyzed (Participants) | 410 | 192
mcg/mL | 9.17 [8.40 to 10.02] | 8.22 [7.17 to 9.41]

14. Primary Outcome: Antibody Response to S. Pneumoniae Serotype 9V - Geometric Mean Titer
Description: Postvaccination observed Geometric Mean Titer of antibody to S. Pneumoniae serotype 9V
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Group 1 - ProQuad™ + PREVNAR™ | Group 2 - PREVNAR™ Followed by ProQuad™
Number analyzed (Participants) | 409 | 193
mcg/mL | 2.98 [2.76 to 3.21] | 2.71 [2.44 to 3.02]

15. Primary Outcome: Antibody Response to S. Pneumoniae Serotype 14 - Geometric Mean Titer
Description: Postvaccination observed Geometric Mean Titer of antibody to S. Pneumoniae serotype 14
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Group 1 - ProQuad™ + PREVNAR™ | Group 2 - PREVNAR™ Followed by ProQuad™
Number analyzed (Participants) | 408 | 193
mcg/mL | 6.88 [6.32 to 7.48] | 5.61 [4.95 to 6.36]

16. Primary Outcome: Antibody Response to S. Pneumoniae Serotype 18C - Geometric Mean Titer
Description: Postvaccination observed Geometric Mean Titer of antibody to S. Pneumoniae serotype 18C
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Group 1 - ProQuad™ + PREVNAR™ | Group 2 - PREVNAR™ Followed by ProQuad™
Number analyzed (Participants) | 408 | 193
mcg/mL | 2.35 [2.14 to 2.58] | 2.23 [1.96 to 2.55]

17. Primary Outcome: Antibody Response to S. Pneumoniae Serotype 19F - Geometric Mean Titer
Description: Postvaccination observed Geometric Mean Titer of antibody to S. Pneumoniae serotype 19F
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Group 1 - ProQuad™ + PREVNAR™ | Group 2 - PREVNAR™ Followed by ProQuad™
Number analyzed (Participants) | 408 | 192
mcg/mL | 3.59 [3.31 to 3.91] | 3.22 [2.85 to 3.64]

18. Primary Outcome: Antibody Response to S. Pneumoniae Serotype 23F - Geometric Mean Titer
Description: Postvaccination observed Geometric Mean Titer of antibody to S. Pneumoniae serotype 23F
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Group 1 - ProQuad™ + PREVNAR™ | Group 2 - PREVNAR™ Followed by ProQuad™
Number analyzed (Participants) | 413 | 197
mcg/mL | 4.24 [3.85 to 4.67] | 3.71 [3.16 to 4.36]

ADVERSE EVENTS:
Time Frame: 28 days post-dose
Description: The number of participants listed as "at risk" is the number of participants with follow-up.
Groups:
- ProQuad™ + Prevnar™ (After Dose 1): ProQuad™ + Prevnar™ (After Dose 1) includes Days 1 to 28 after the first dose of ProQuad™ (safety follow-up period 1 for Group 1)
- ProQuad™ Alone (After Dose 1): ProQuad™ Alone (After Dose 1) includes Days 1 to 28 after the first dose of ProQuad™ (safety follow-up period 1 for Group 3 and safety follow-up period 2 for Group 2).
- ProQuad™ (After Dose 2): ProQuad™ (After Dose 2) includes Days 1 to 28 after the second dose of ProQuad™ (safety follow-up period 3 for Group 1, Group 2, and Group 3).
Arm/Group | ProQuad™ + Prevnar™ (After Dose 1) | ProQuad™ Alone (After Dose 1) | ProQuad™ (After Dose 2)
Serious Adverse Events (participants affected / at risk) | 4/498 | 3/495 | 0/910
Other Adverse Events (participants affected / at risk) | 367/498 | 311/495 | 499/910
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ProQuad™ + Prevnar™ (After Dose 1) (N=498) | ProQuad™ Alone (After Dose 1) (N=495) | ProQuad™ (After Dose 2) (N=910)
Pneumonia (Infections and infestations) | 2 | 0 | 0
Pneumonia Viral (Infections and infestations) | 1 | 0 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Croup Infectious (Infections and infestations) | 0 | 1 | 0
Febrile Convulsion (Nervous system disorders) | 0 | 1 | 0
Neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | ProQuad™ + Prevnar™ (After Dose 1) (N=498) | ProQuad™ Alone (After Dose 1) (N=495) | ProQuad™ (After Dose 2) (N=910)
Conjunctivitis (Eye disorders) | 10 | 6 | 7
Diarrhoea (Gastrointestinal disorders) | 31 | 16 | 25
Vomiting (Gastrointestinal disorders) | 16 | 16 | 25
Irritability (General disorders) | 27 | 16 | 13
Pyrexia (General disorders) | 112 | 109 | 138
Gastroenteritis (Infections and infestations) | 9 | 12 | 15
Nasopharyngitis (Infections and infestations) | 7 | 21 | 40
Otitis Media (Infections and infestations) | 28 | 32 | 57
Otitis Media Acute (Infections and infestations) | 13 | 2 | 7
Pharyngitis (Infections and infestations) | 5 | 2 | 6
Pneumonia (Infections and infestations) | 5 | 2 | 4
Sinusitis (Infections and infestations) | 6 | 3 | 11
Upper Respiratory Tract Infection (Immune system disorders) | 59 | 46 | 94
Viral Infection (Infections and infestations) | 10 | 10 | 12
Viral Rash (Infections and infestations) | 7 | 5 | 5
Arthropod Bite (Infections and infestations) | 2 | 6 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 14 | 39
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 6 | 11
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 21 | 16 | 36
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 26 | 11 | 19
Eczema (Skin and subcutaneous tissue disorders) | 7 | 4 | 11
Rash (Skin and subcutaneous tissue disorders) | 23 | 19 | 14
Rash Morbilliform (Skin and subcutaneous tissue disorders) | 27 | 24 | 15
Rash Vesicular (Skin and subcutaneous tissue disorders) | 10 | 6 | 4
Injection Site Bruising (Prevnar Injection-site) (Skin and subcutaneous tissue disorders) | 8 | 0/0 | 0/0
Injection Site Erythema (Prevnar Injection-site) (Skin and subcutaneous tissue disorders) | 106 | 0/0 | 0/0
Injection Site Pain (Prevnar Injection-site) (Skin and subcutaneous tissue disorders) | 157 | 0/0 | 0/0
Injection Site Rash (Prevnar Injection-site) (Skin and subcutaneous tissue disorders) | 5 | 0/0 | 0/0
Injection Site Swelling (Prevnar Injection-site) (Skin and subcutaneous tissue disorders) | 92 | 0/0 | 0/0
Injection Site Bruising (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 10 | 8 | 3
Injection Site Erythema (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 69 | 67 | 153
Injection Site Pain (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 125 | 127 | 163
Injection Site Rash (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 6 | 12 | 9
Injection Site Swelling (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 58 | 54 | 118

LIMITATIONS AND CAVEATS:
One subject (Group 3-ProQuad™ followed by PREVNAR™) was diagnosed (Day 8) with Stage IV neuroblastoma (considered not related to study vaccine by investigator) and discontinued from the study. Subject died (Day 218) due to neuroblastoma.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.